CLINICAL TRIAL: NCT01958619
Title: Open Label Pharmacokinetic Study of OZ439 and Piperaquine Following Administration of OZ439+TPGS Granules for Oral Suspension Alone or With Either Piperaquine Phosphate Tablets or Granules for Oral Solution in the Fasted State in Healthy Volunteers
Brief Title: Open Label Pharmacokinetic Study of OZ439 and Piperaquine on Administration of OZ439+TPGS Granules for Oral Suspension Alone or With Either Piperaquine Phosphate Tablets or Granules for Oral Solution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMV_OZ439_13_004; 2013-003409-25 (EudraCT Number)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2015-04-21 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Malaria
Keywords: open label; healthy volunteers; pharmacokinetic; parallel group
MeSH Terms: conditions — Malaria | interventions — artefenomel; tocophersolan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A: 1440mg PQP tablets & 800mg OZ439 + TPGS (Experimental): Piperaquine phosphate tablets (1440mg) and OZ439 (800mg) + TPGS granules for oral suspension under fasted conditions.
  Interventions: Drug: 1440mg PQP tablets; Drug: 800mg OZ439 + TPGS
- Treatment B: 960mg PQP tablets & 800mg OZ439 + TPGS (Experimental): Piperaquine phosphate tablets (960mg) and OZ439 (800mg) + TPGS granules for oral suspension under fasted conditions.
  Interventions: Drug: 960mg PQP tablets; Drug: 800mg OZ439 + TPGS
- Treatment C: 960mg PQP granules & 800mg OZ439 + TPGS (Experimental): Piperaquine phosphate granules for oral solution (960mg) and OZ439 (800mg) + TPGS granules for oral suspension under fasted conditions.
  Interventions: Drug: 800mg OZ439 + TPGS; Drug: 960mg PQP granules
- Treatment D: 800mg OZ439 + TPGS (Experimental): OZ439 (800mg) + TPGS granules for oral suspension under fasted conditions.
  Interventions: Drug: 800mg OZ439 + TPGS

INTERVENTIONS:
Drug: 1440mg PQP tablets — Piperaquine phosphate tablets (1440mg)
  Arms: Treatment A: 1440mg PQP tablets & 800mg OZ439 + TPGS
Drug: 960mg PQP tablets — Piperaquine phosphate tablets (960mg)
  Arms: Treatment B: 960mg PQP tablets & 800mg OZ439 + TPGS
Drug: 800mg OZ439 + TPGS — OZ439 (800mg) + TPGS granules for oral suspension
Drug: 960mg PQP granules — Piperaquine phosphate granules for oral solution (960mg)
  Arms: Treatment C: 960mg PQP granules & 800mg OZ439 + TPGS

SUMMARY:
A healthy volunteer study to characterise the exposure of the two study medications, following administration of OZ439 + TPGS granules with piperaquine phosphate granules (intended for children) and with piperaquine phosphate tablets (intended for adults). Ideally, to confirm the exposure demonstrated in an earlier bioavailability study.

DETAILED DESCRIPTION:
A Phase 1 open label parallel group, four arm study conducted in healthy male and female subject aged 18 to 55 years of age. Subjects will receive either treatment A, B, C or D as described below:

* Treatment A: 1440 mg PQP tablets and 800 mg OZ439 + TPGS granules for oral suspension
* Treatment B: 960 mg PQP tablets and 800 mg OZ439 + TPGS granules for oral suspension
* Treatment C: 960 mg PQP granules for oral solution and 800 mg OZ439 + TPGS granules for oral suspension
* Treatment D: 800 mg OZ439 + TPGS granules for oral suspension

ELIGIBILITY:
Inclusion Criteria:

* healthy, male or female, any race aged 18-55 years at screening
* body mass index of 18-30kg/m2 inclusive; and a total body weight >50kg and up to 100kg at screening
* Females must have negative pregnancy test at screening, be non-lactating and of non-childbearing potential confirmed by:

  * natural (spontaneous) post-menopausal defined as amenorrheic for 12 months without an alternative medical cause with a screening FSH level >25IU/L for post menopause
  * irreversible surgical sterilisation by bilateral oophorectomy or bilateral salpingectomy but not tubal ligation (with or without hysterectomy) at least six months ago
* Must agree to use acceptable methods of contraception Males must use acceptable methods of contraception if the male subject's partner could become pregnant from the time of the first administration of treatment or study medication until 3 months following administration of the last dose of study medication

One of the following acceptable methods of contraception must be used:

* Condom & occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository)
* Surgical sterilisation (vasectomy with documentation of azoospermia) and a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps] used with spermicidal foam/gel/film/cream/suppository)
* Female partner uses oral contraceptives (combination oestrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method (as above)
* Female partner uses medically prescribed topically-applied transdermal contraceptive patch and a barrier method (as above)
* Female partner has had documented tubal ligation (sterilization). In addition, a barrier method (as above) must be used
* Female partner has had documented placement of an intrauterine device or system and the use of a barrier method (as above)
* True abstinence: when in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Abstinent subjects must agree use one of the above-mentioned contraceptive methods, if sexual relationships start during the study or up to 90 days after the last dose of study drug

  * Subjects should not donate egg and sperm from the time of administration of study medication until 3 months after study medication
  * Must be capable of understanding and complying with the requirements of the protocol and must have signed the informed consent form prior to undergoing any study-related procedures

Exclusion Criteria:

* Male subjects with female partner(s) who is (are) pregnant or lactating from the time of the administration of study medication
* Has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion
* History of allergic reaction to artemisinin-based compounds, 4-aminoquinolines such as piperaquine or any other clinically relevant allergy to drugs or food
* Any clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at screening or on admission
* History or current evidence of any clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal (excluding appendectomy and cholecystectomy), haematological, endocrinological, immunological, metabolic, neurological, oncological, psychiatric, urological or other disease, or current infection
* History of post-antibiotic colitis
* Electrocardiogram abnormalities in the 12-lead Electrocardiogram (at screening) and/or 24-hour Holter Electrocardiogram (at screening) which in the opinion of the Investigator is clinically relevant or will interfere with the ECG analysis
* History of clinically significant Electrocardiogram abnormalities, or any of the following abnormalities at screening or on admission:

  * PR >200ms
  * QRS complex >120ms
  * QTcB or QTcF >450ms or shortened QTcB or QTcF less than 340ms for males and females or family history of long QT syndrome or sudden death
  * Any degree of heart block (such as first, second or third degree atrioventricular block, incomplete, full or intermittent bundle branch block)
  * Abnormal T wave morphology / prominent U waves
* Positive results in any of the serology tests for Hepatitis B Surface Antigen, anti Hepatitis core antibody, Hepatitis C antibodies, and HIV 1 and 2 antibodies
* Confirmed positive results from urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates, and methadone) or from the alcohol breath test at screening and admission
* History or clinical evidence of alcohol abuse, or any recreational drug abuse within the 2 years of screening
* Mentally handicapped
* Participation in a drug trial within 90 days of drug administration
* Use of ANY prescription or over the counter medications, within 3 weeks of study medication administration, or vitamins or herbal supplements within 2 weeks of administration of the study drug, unless prior approval is granted. Intermittent use of paracetamol at doses of up to 2g/day is permitted
* Use of moderate/strong inhibitors and/or inducers of CYP450 in 4 weeks of drug administration (or at least 5 half-lives of the compound whichever is the longer)
* Veins unsuitable for intravenous puncture or cannulation on either arm (veins difficult to locate, access or puncture, or veins with a tendency to rupture during or after puncture)
* Transaminases, bilirubin, serum potassium outside normal range at screening or admission
* Haemoglobin < lower limit of normal at screening or admission
* Donation of >500mL blood in 90 days prior to drug administration
* Must be non-smoker for at least three months before screening. "Tobacco use" includes smoking and the use of snuff and chewing tobacco, and other nicotine containing products. May not use any non-nicotine containing smoking cessation aids, e.g. varenicline, for at least three months before screening
* Any consumption of grapefruit, Seville oranges, wild grapes, black mulberries, pomegranates as fruit juice, marmalade or as a raw fruit within 7 days prior to dosing of study drug and throughout the study
* Any circumstances or conditions, which may affect full participation in the trial or compliance with the protocol
* Legal incapacity or limited legal capacity at screening
* Vegetarians, vegans or any dietary restrictions conflicting with the study standardised menus

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD FRCA FFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd., Croydon, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment A: 1440mg PQP Tablets & 800mg OZ439 + TPGS | Treatment B: 960mg PQP Tablets & 800mg OZ439 + TPGS | Treatment C: 960mg PQP Granules & 800mg OZ439 + TPGS | Treatment D: 800mg OZ439 + TPGS
Started | 15 | 14 | 14 | 12
Completed | 13 | 14 | 13 | 12
Not Completed | 2 | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one single dose of OZ439 or Piperaquine
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A: 1440mg PQP Tablets & 800mg OZ439 + TPGS | Treatment B: 960mg PQP Tablets & 800mg OZ439 + TPGS | Treatment C: 960mg PQP Granules & 800mg OZ439 + TPGS | Treatment D: 800mg OZ439 + TPGS | Total
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (9.40) | 31.8 (9.70) | 26.9 (5.66) | 28.6 (9.54) | 28.5 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 2
  Male | 14 | 14 | 14 | 11 | 53
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 14 | 14 | 12 | 55

OUTCOME MEASURES:

1. Primary Outcome: OZ439 Cmax
Description: OZ439 observed maximum drug plasma concentration
Time Frame: Days 1 pre-dose and post-dose at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16 and 24 hours (Day 2), and, 48 (Day 3), 72 (Day 4), 96 (Day 5) and 168 (Day 8) hours post-dose. Sampling will also be done on Day 11, 15, 29 and 43.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: 1440mg PQP Tablets & 800mg OZ439 + TPGS | Treatment B: 960mg PQP Tablets & 800mg OZ439 + TPGS | Treatment C: 960mg PQP Granules & 800mg OZ439 + TPGS | Treatment D: 800mg OZ439 + TPGS
Number analyzed (Participants) | 13 | 14 | 13 | 12
ng/mL | 1300 (34.6) | 1490 (37.9) | 1240 (29.2) | 1120 (48.6)

2. Primary Outcome: OZ439 AUC0-∞
Description: OZ439 Area under plasma concentration time curve from time zero extrapolated to infinity.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: 1440mg PQP Tablets & 800mg OZ439 + TPGS | Treatment B: 960mg PQP Tablets & 800mg OZ439 + TPGS | Treatment C: 960mg PQP Granules & 800mg OZ439 + TPGS | Treatment D: 800mg OZ439 + TPGS
Number analyzed (Participants) | 13 | 14 | 13 | 12
ng*h/mL | 15000 (26.3) | 16100 (35.7) | 14100 (35.9) | 13400 (53.7)

3. Secondary Outcome: Piperaquine Cmax
Description: Piperaquine Observed maximum drug plasma concentration
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: 1440mg PQP Tablets & 800mg OZ439 + TPGS | Treatment B: 960mg PQP Tablets & 800mg OZ439 + TPGS | Treatment C: 960mg PQP Granules & 800mg OZ439 + TPGS
Number analyzed (Participants) | 13 | 14 | 13
ng/mL | 249 (94.3) | 113 (100.9) | 112 (68.7)

4. Secondary Outcome: Piperaquine AUC0-∞
Description: Piperaquine Area under plasma concentration time curve from time zero extrapolated to infinity.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: 1440mg PQP Tablets & 800mg OZ439 + TPGS | Treatment B: 960mg PQP Tablets & 800mg OZ439 + TPGS | Treatment C: 960mg PQP Granules & 800mg OZ439 + TPGS
Number analyzed (Participants) | 13 | 14 | 13
ng*h/mL | 18300 (39.3) | 12400 (43.2) | 12100 (42.1)

ADVERSE EVENTS:
Time Frame: Up to Day 50 post-dose.
Description: All 55 subjects received one dose of OZ439 alone or in combination with PQP were included in the safety analysis population
Arm/Group | Treatment A: 1440mg PQP Tablets & 800mg OZ439 + TPGS | Treatment B: 960mg PQP Tablets & 800mg OZ439 + TPGS | Treatment C: 960mg PQP Granules & 800mg OZ439 + TPGS | Treatment D: 800mg OZ439 + TPGS
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 8/15 | 5/14 | 8/14 | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: 1440mg PQP Tablets & 800mg OZ439 + TPGS (N=15) | Treatment B: 960mg PQP Tablets & 800mg OZ439 + TPGS (N=14) | Treatment C: 960mg PQP Granules & 800mg OZ439 + TPGS (N=14) | Treatment D: 800mg OZ439 + TPGS (N=12)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (3) | 5 (5) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling Hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion of the study, the Investigator may prepare a joint publication with MMV. The Investigator must undertake not to submit any part of the individual data from this protocol for publication without prior consent of MMV at a mutually agreed time. The confidentiality obligation applies to all personnel involved at the investigational site.